CLINICAL TRIAL: NCT02507050
Title: Can Ivabradine Attenuate Post-revascularisation Microcirculatory Dysfunction in Flow Limiting Coronary Artery Disease?
Brief Title: Ivabradine and Post-revascularisation Microcirculatory Dysfunction
Acronym: MICRO-PCI
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding not yet achieved
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1060
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Coronary Artery Disease; Angina
Keywords: Ivabradine; Microvascular dysfunction; PCI; Procedural related myocardial injury; IMR; Index of Microvascular Resistance
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris | interventions — Ivabradine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Patients randomised to stop beta blockers and start Ivabradine. Initial dose of 5mg BD, titrated to 7.5mg BD if possible.
  Interventions: Drug: Ivabradine
- Standard therapy (No Intervention): Bisoprolol given as standard beta blocker treatment i.e. Bisoprolol (maximum dose 10mg OD).

INTERVENTIONS:
Drug: Ivabradine — To start Ivabradine 6 weeks prior to PCI.
  Other Names: Procoralan
  Arms: Intervention

SUMMARY:
The aim of the study is to test whether, in patients with angina and flow limiting epicardial coronary artery disease, pre-treatment with Ivabradine, as opposed to beta blockers, will reduce post percutaneous coronary intervention induced microvascular dysfunction.

DETAILED DESCRIPTION:
We will be recruiting patients with stable angina referred for percutaneous intervention (PCI) due to flow limiting coronary artery disease. All patients will be on an existing beta blocker prescription (standard first line angina therapy). Our hypothesis is that Ivabradine will attenuate microvascular dysfunction post PCI when compared to standard beta-blocker pre-treatment. We intend to test this in a randomised, open-label parallel arm study with a direct comparison between Ivabradine and beta-blockers (standard therapy). Patients will be randomised to receive either Ivabradine (and stop beta blockers) or continue beta blockers for 6 weeks prior to the PCI procedure. The primary endpoint will be IMR (index of microvascular resistance) post PCI, as a marker of microvascular dysfunction and procedural related myocardial injury. IMR is a potent marker of adverse outcome in STEMI patients and in ACS after PCI. Although this has yet to be assessed in the elective setting, a reduction in IMR with Ivabradine may indicate a potential to improve outcomes and lessen iatrogenic microvascular dysfunction post PCI. IMR is assessed using thermodilution catheters placed distal to the coronary stenosis and by producing hyperaemia. To assess the medium term effects on the microcirculation post PCI all patients will have a stress perfusion cardiac MRI 12 weeks post procedure. The secondary endpoint will be proportion of patients with coronary flow reserve (CFR) <2.0 in PCI territory (regional myocardial blood flow at hyperaemia by intravenous adenosine infusion compared to rest). We will also be assessing CFI (collateral flow index), as promotion of the collateral system is one method by which Ivabradine may lessen procedural related myocardial injury, and ΔIMR as the difference between IMR pre and post-PCI.

The measurement of cardiac troponins and use of cardiac MRI will facilitate the identification of peri-procedural myocardial injury and procedural related myocardial infarction as further secondary end points. The Seattle Angina Questionnaire will be used at 3 intervals to assess symptoms throughout the study. The total study length for each patient will be 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms of Angina Pectoris
2. Angiographic evidence of epicardial coronary artery stenosis referred for PCI
3. Flow limiting lesion (Fractional Flow Reserve ≤0.80) in one of following locations (as defined in SYNTAX trial89):

   1. Proximal or mid left anterior descending artery (LAD)
   2. Proximal or mid dominant right coronary artery (RCA)
   3. Proximal left circumflex artery (LCx) or 1ST Obtuse marginal Vessel
4. Existing beta blocker prescription
5. Echocardiogram performed within preceding 12 months
6. Patient consent

Exclusion Criteria:

1. Previous myocardial infarction (MI) in target vessel myocardial territory or any MI in preceding 12 months (defined by patient history, ECG changes and evidence of regional wall motion abnormalities on echocardiography)
2. FFR>0.80 in target vessel at time of procedure
3. Requirement for Multi-vessel intervention in a single procedure
4. Any chronic total occlusion (100% epicardial occlusion) on angiography
5. Distal coronary artery stenosis or that affecting non-dominant RCA
6. Heart Rate <60 bpm at inclusion (assessed by 12 lead ECG after minimum 10 minutes rest period)
7. Any rhythm other than sinus rhythm
8. Sick sinus syndrome or high grade atrio-ventricular block
9. Permanent Pacemaker in situ
10. Congenital QT Syndrome
11. Intolerance or allergy to beta-blockers
12. Intolerance to Ivabradine
13. Additional (other than angina pectoris) indication for beta-blocker treatment e.g. ventricular tachycardia
14. Concurrent required use of rate-limiting drugs other than beta-blockers
15. The necessity of combination therapy with Ivabradine and bisoprolol to achieve heart rate control
16. Contraindication to Magnetic Resonance Imaging or IV adenosine
17. Severe impairment of renal function (eGFR<30ml/min)
18. Severe Liver Disease (Any worse than Grade A by Child-Pugh Classification)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
IMR (Index of Microvascular Resistance) | Immediately after PCI
  Invasive marker of microvascular dysfunction

SECONDARY OUTCOMES:
Peri-procedural Troponin Release | 3 hours after PCI
  Rise in high sensitivity troponin 3 hours after PCI
CFI pre-revascularisation | Immediately prior to PCI
  Collateral flow index is an invasively measured marker of collateral blood flow- to be measured prior to PCI
Symptomatic Improvement (Seattle Angina Questionnaire) | 18 weeks
  Seattle Angina Questionnaire assessed at 18 weeks after starting treatment (12 weeks after PCI) and compared to baseline scores.
Coronary Flow Reserve | 12 weeks
  Coronary Flow Reserve measured in target vessel on MRI at 12 weeks after PCI

CONTACTS AND LOCATIONS:
Overall Officials: Aleem Khand, MBChB MD, Principal Investigator — Liverpool Heart and Chest Hospital
Locations (1):
- Liverpool Heart and Chest Hospital, Liverpool, United Kingdom